CLINICAL TRIAL: NCT00411229
Title: A Phase III Study Comparing Adjuvant Chemotherapy Consisting of Capecitabine/Oxaliplatin vs Surgery Alone in Patients With Stage II (T1N2, T2N1, T3N0), IIIa (T2N2, T3N1, T4NO), and IIIb (T3N2) Gastric Adenocarcinoma
Brief Title: Capecitabine and Oxaliplatin Adjuvant Study in Stomach Cancer
Acronym: CLASSIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L_9570; M017527
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (2):
- 1 (Active Comparator): Capecitabine + Oxalipatin
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- 2 (No Intervention)

INTERVENTIONS:
Drug: Capecitabine — 1,000 mg/m² twice daily. Film coated tablets of 500 mg, 150mg.
  Arms: 1
Drug: Oxaliplatin — IV infusion, 130mg/m²
  Arms: 1

SUMMARY:
Primary:

* To demonstrate that capecitabine/oxaliplatin as adjuvant chemotherapy is superior to observation alone in terms of 3 year disease-free survival (DFS) rate in chemotherapy-naïve patients who underwent potentially curative resection for gastric cancer.

Secondary:

* To compare the overall survival of surgery and capecitabine/ oxaliplatin as adjuvant therapy versus surgery alone. To evaluate the safety profile of capecitabine/oxaliplatin adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients
* Karnofsky performance status of ≥70 %.
* Histologically confirmed gastric adenocarcinoma, staged pathologically, stage II (T2N1, T1N2, T3N0), IIIa (T3N1, T2N2, T4N0), and IIIb (T3N2). At least 15 examined lymph nodes are required to ensure the adequate TNM (Tumor Nodes Metastases classification.
* Patients who underwent curative D2 lymphadenectomy resection for gastric cancer with no macroscopic or microscopic evidence for remaining tumor, who can be randomized to either study arm within 6 weeks after surgery.

Exclusion Criteria:

* Pregnant or lactating women.
* Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Any evidence of metastatic disease (including presence of tumor cells in the ascites).
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
* Known peripheral neuropathy ≥ CTCAEv3 grade 1 (Common Terminology for Adverse Events). Absence of deep tendon reflexes as the sole neurologic abnormality does not render the patient ineligible.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Moderate or severe renal impairment [creatinine clearance equal to or below 50 ml/min (calculated according to Cockroft and Gault)], or serum creatinine > 1.5 x upper limit of normal (ULN).
* Any of the following laboratory values:

  * Absolute neutrophil count (ANC) < 1.5 x 109/L
  * Platelet count < 100 x 109/L
  * Total bilirubin > 1.5 x ULN
  * ALAT, ASAT > 2.5 x ULN
  * Alkaline phosphatase > 2.5 x ULN.
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented dihydropyrimidine dehydrogenase (DPD) deficiency) or patients with known DPD deficiency.
* Hypersensitivity to platinum compounds or any of the components of the study medications.
* Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before randomization.
* Blood transfusions or growth factors to aid hematologic recovery within 2 weeks prior to study treatment start.
* Requirement for concurrent use of the antiviral agent sorivudine (antiviral) or chemically related analogues, such as brivudine.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2006-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Recurrence of the original cancer | From the beginning to end of the study
Development of a new gastric cancer | From beginning to end of study
Death due to any cause | From the beginning to the end of study
Adverse events | From beginning to end of study
Clinical laboratory tests | From beginning to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis, Beijing, China
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Taipei, Taiwan

REFERENCES:
- [Derived] Cheong JH, Yang HK, Kim H, Kim WH, Kim YW, Kook MC, Park YK, Kim HH, Lee HS, Lee KH, Gu MJ, Kim HY, Lee J, Choi SH, Hong S, Kim JW, Choi YY, Hyung WJ, Jang E, Kim H, Huh YM, Noh SH. Predictive test for chemotherapy response in resectable gastric cancer: a multi-cohort, retrospective analysis. Lancet Oncol. 2018 May;19(5):629-638. doi: 10.1016/S1470-2045(18)30108-6. Epub 2018 Mar 19. PMID 29567071
- [Derived] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Derived] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517